CLINICAL TRIAL: NCT04826744
Title: Frequency of Palpebral Involvement in Adult Atopic Dermatitis, in a Cohort of Patients From Lille and Rouen (France) ; a Multicenter Prospective Study
Brief Title: Frequency of Palpebral Involvement in Adult With Atopic Dermatitis
Acronym: PAUPIAD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_15; 2020-A02373-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-03-16; First posted 2021-04-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic eczema; palpebral dermatitis; patch-testing; ophthalmology; allergology; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with palpebral involvement of atopic dermatitis
  Interventions: Other: Standard dermatology consultation

INTERVENTIONS:
Other: Standard dermatology consultation — with clinical examination, score filling such as SCORAD and DLQI
  * Standard Allergy consultation, with clinical examination, research of atopic or allergic personal and familial history
  * Allergy skin testing: patch tests with the Standard European Battery and with some products bring by the patient if necessary, skin prick tests with aero allergens. Two reading of the patch tests will be performed, at H48 and H72.
  * ophthalmologic consultation with slit lamp examination and OSDI (self questionnaire)

SUMMARY:
Atopic dermatitis is a common inflammatory skin disease, resulting from genetical, immunological and environmental factors. Head and neck are among the most frequent involved areas, almost 50% in adult patients according to most publications. Palpebral involvement is also common and a source of major quality of life impairment for patients.

However, the real frequency of this palpebral involvement is unknown, only estimated about 20% in few studies. The treatment of this location remains difficult, regarding to the thickness of palpebral skin and proximity of the eye.

To our knowledge, no prospective studies about allergological skin tests (such as patch-tests) in atopic patients with palpebral involvement had been conducted.

Finally, atopic dermatitis is frequently associated with ophthalmological diseases such as conjunctivitis, keratoconus or cataract, which belong to the minor criteria of Hanifin and Rakja classification.

A better knowledge of the atopic dermatitis palpebral involvement and the associated factors seems to be needed to improve the treatment and the quality of life of patients

ELIGIBILITY:
Inclusion Criteria:

* Atopic Dermatitis according to the revised Hanifin and Rakja criteria (UK Working Party)
* Oral consent
* Valid social insurance

Exclusion Criteria:

* Personal history of uncontrolled asthma
* No social insurance
* Protective measures
* Age under 18
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with atopic dermatitis. Systematic inclusion of out-patients and in-patients of the University Hospital of Lille and Rouen, but also patients from liberal physicians (dermatologists and allergists) in Lille and Rouen
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ratio of palpebral involvement in adult atopic dermatitis patients, regardless the severity of the disease | At Baseline, the initial consultation of dermatology

SECONDARY OUTCOMES:
Clinical description of the palpebral involvement : acute eczema or chronic eczema | At Baseline, the initial consultation of dermatology
Potential factors associated with palpebral involvement of the atopic dermatitis (socio-demographics factors, clinical factors, comorbidities, treatment, severity …) | At Baseline, (the initial consultation of dermatology ) and at 3 months during the consultation of allergology
Rate of relevant contact sensitization according to the skin testing and the clinical manifestations | At 3 months, at the time of the reading of the tests either at 48 hours and 72 hours
Description of the sensitization profile | At 3 months, at the time of the reading of the tests either at 48 hours and 72 hours
Association between allergic sensitization and severity of the atopic dermatitis | At 3 months, at the time of the reading of the tests either at 48 hours and 72 hours
Rate of ophthalmologic comorbidities in association with palpebral involvement of the atopic dermatitis | At 3 months during the time of the ophthalmologic consultation
Clinical description of the ophthalmologic involvement and OSDI scoring | At 3 months during the time of the ophthalmologic consultation
Association between allergic sensitization and ophthalmologic involvement | At 3 months, at the time of the reading of the tests either at 48 hours and 72 hours
Association between ophthalmologic involvement and severity of the atopic dermatitis | At 3 months, at the time of the reading of the tests either at 48 hours and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Staumont-Salle, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hop Claude Huriez Chu Lille, Lille
  - Hopital Charles Nicolle Chu Rouen, Rouen